CLINICAL TRIAL: NCT04874727
Title: Reduction of Volumetric and AP Measurements of the Airway in Pseudo-sleep Supine Position vs Standard 3D Cone Beam Computed Tomography on Patients With Sleep Apnea
Brief Title: Comparison of Standing Versus Supine 3D Cone Beam Computed Tomography in Patient With Obstructive Sleep Apnea
Acronym: OSA
Status: Completed | Type: Observational
Sponsor: Manhattan Beach Orthodontics (Other)
Responsible Party: Principal Investigator, Dr. Maryam Bakhtiyari, Dentist, Owner, Manhattan Beach Orthodontics
Other Study IDs: 0002
Record Dates: First submitted 2021-01-18; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: OSA; Sleep Apnea
Keywords: tomography; CBCT; Cone-beam computerized tomography; obstructive sleep apnea; airway volume; anterior-posterior measurement
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: The five or six individual patients enrolled are the members of the sole group, the study population. These individuals all have been diagnosed with obstructive sleep apnea and have take a Cone-beam CT scan with and without the new bite technique.
  Interventions: Procedure: Mandible slacked and captured with Correct Plus™ Impression Material Superfast

INTERVENTIONS:
Procedure: Mandible slacked and captured with Correct Plus™ Impression Material Superfast — In order to simulate the supine position, patients are placed in a supine position (180 degrees) in a dental exam chair, and asked to relax their lower jaw, allowing it to drop back, simulating their jaw falling back while sleeping. That bite is then captured with a Correct Plus™ Impression Material Superfast. Once the bite material hardens, it locks the bite in place. The patient then stands upright, and CBCT is taken standing while the jaw placement is still pseudo sleep-supine, supported by the bite material.

SUMMARY:
The anatomical changes of the upper airway in a standing vs pseudo-supine position using Carestream Orthodontic Imaging (Volumetric) and Carestream Orthodontic Imaging module (AP measurements) of the patient's airway respectively, have been taken and the obtained results compared. In order to simulate the supine position, patients are placed in a supine position (180 degrees) in a dental exam chair, and asked to relax their lower jaw, allowing it to drop back, simulating their jaw falling back while sleeping. That bite is then captured with a Correct Plus™ Impression Material Superfast. Once the bite material hardens, it locks the bite in place. The patient then stands upright, and CBCT is taken standing while the jaw placement is still pseudo sleep-supine, supported by the bite material.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a patient of Dr. Maryam Bakhtiyari's orthodontic practice
* Participant must have a diagnosis of obstructive sleep apnea
* Participant must have an invitation to join research study from Dr. Bakhtiyari

Exclusion Criteria:

* Participant cannot have a history of serious dental trauma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population was selected from the patient pool of Dr. Maryam Bakhtiyari. They are individuals with diagnoses of OSA and consented to taking two x-rays and enrolling into this study.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
3D volumetric airway measurement | through study completion, an average of 1 year
  Investigators will measure and compare the 3D volumetric airway of the x-ray both with and without the pseudo-supine technique. This will be done on the computer using Carestream Orthodontic Imaging.
2D Anterior-Posterior airway Measurement | through study completion, an average of 1 year
  Investigators will measure and compare the 2D anterior-posterior airway of the x-ray both with and without the pseudo-supine technique. This will be done on the computer using the Carestream Orthodontic Imaging module.

CONTACTS AND LOCATIONS:
Locations (1):
- Manhattan Beach Orthodontics, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No